CLINICAL TRIAL: NCT04844931
Title: Randomized Comparison of Combined Remote Ischemic Conditioning and Local Postconditioning Compared to Standard Treatment in High-risk ST-elevation Myocardial Infarction Patients
Brief Title: Remote Ischemic Conditioning With Local Ischemic Postconditioning in High-Risk ST-elevation Myocardial Infarction
Acronym: RIP-HIGH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0089
Record Dates: First submitted 2021-03-31; First posted 2021-04-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: remote ischemic conditioning; local ischemic postconditioning; percutaneous coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: patients will be randomized to one of the two groups in a 1:1 ratio stratified by center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC + PostC in addition to standard treatment (Experimental): RIC by arm ischemia initiated on hospital admission plus local PostC by re-inflating the angioplasty balloon after re-opening the infarct-related artery in addition to standard treatment.
  Interventions: Procedure: RIC + PostC + Standard PCI
- Standard treatment (Active Comparator)
  Interventions: Procedure: Standard PCI

INTERVENTIONS:
Procedure: RIC + PostC + Standard PCI — RIC by arm ischemia initiated on hospital admission plus local PostC by re-inflating the angioplasty balloon after re-opening the infarct-related artery
  Arms: RIC + PostC in addition to standard treatment
Procedure: Standard PCI — Standard PCI
  Arms: Standard treatment

SUMMARY:
The RIP-HIGH trial is a two-arm randomized controlled trial aiming to compare the impact of combined remote ischemic conditioning (RIP) and local ischemic postconditioning (PostC) vs. standard of care on clinical outcome in high-risk ST-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Coronary reperfusion by percutaneous coronary intervention is mandatory to salvage ischemic myocardium and to reduce definite infarct size. However, reperfusion itself also causes irreversible myocardial damage - a phenomenon described as reperfusion injury. Reduction of ischemic and reperfusion injury by ischemic conditioning has been identified as a potential target to reduce myocardial damage.

Remote ischemic conditioning and local ischemic postconditioning might be in particular of clinical benefit in higher risk STEMI patients with Killip class ≥2, where mortality rates are high.

The Remote Ischemic Conditioning with Local Ischemic Postconditioning in High-Risk ST-elevation myocardial infarction patients (RIP-HIGH) trial is a two-arm randomized controlled trial aiming to compare the impact of combined remote ischemic conditioning and local ischemic postconditioning vs. standard of care on clinical outcome in high-risk ST-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain lasting <12 h
* ST-elevation at the J-point in two contiguous leads of ≥2 mm in men ≥40 years, ≥2.5 mm in men <40 years and ≥1.5 mm in women (regardless of age) in V2-V3 and/or ≥1 mm in all other leads (52).
* New or presumed new left bundle branch block or right bundle branch block.
* Killip class ≥II on hospital admission or requirement of diuretics because of clinical congestion.
* Written informed consent.

Exclusion Criteria:

* Killip class I on hospital admission.
* Prior fibrinolysis.
* Conditions precluding use of RIC (i.e. paresis of the upper limb, presence of an arteriovenous shunt).
* Pregnancy.
* Age <18 years.
* Severe co-morbidity with a life expectancy <6 months.
* Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or hospitalization for heart failure (HF) within 12 months after randomization. | 12 months

SECONDARY OUTCOMES:
All-cause mortality at 12 months | 12 months
Hospitalization for heart failure at 12 months | 12 months
Composite of all-cause mortality, HF hospitalization and survived out-of-hospital cardiac arrest at 12 months | 12 months
Cardiovascular mortality at 12 months. | 12 months
Enzymatic infarct size defined as high-sensitivity cardiac troponin T (hs-TnT) levels 72 h after randomization | day 3
Change in N-terminal pro B-type natriuretic peptide (NT-proBNP) levels during admission and 72 h after randomization | day 0, day 3
Thrombolysis in myocardial infarction (TIMI)-flow grade of the culprit vessel post PCI | day 0
Proportion of patients showing complete (≥70%) resolution of ST-segment elevation 60 minutes after reperfusion | day 0
CMR-derived infarct size. | day 2-5
CMR-derived myocardial salvage index | day 2-5
Extent of CMR-derived late microvascular obstruction on day 2-5 after randomization | day 2-5
all-cause mortality, HF hospitalization and survived out-of-hospital cardiac arrest assessed at 5 years via telephone contact. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Prof. Dr., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (11):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Germany (10):
  - Klinikum Links der Weser, Bremen
  - Herzzentrum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Hospital Essen, Essen
  - University Clinic Hamburg-Eppendorf, Hamburg
  - Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen
  - University Heart Center Lübeck - University of Schleswig-Holstein, Lübeck
  - Universitätsmedizin Rostock, Rostock
  - University Hospital Tübingen, Tübingen